CLINICAL TRIAL: NCT01098227
Title: A Prospective Study Measuring Exhaled Nitric Oxide Levels in Infants and Young Children Admitted to the Hospital for Respiratory Syncytial Virus (RSV) or Other Viral Lower Respiratory Tract Infections
Brief Title: Exhaled Nitric Oxide Levels in Infants and Young Children Infected With RSV or Other Viral Infections
Status: Withdrawn | Type: Observational
Why Stopped: The equipment to be used for the study was inoperable and not repairable.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 147914
Record Dates: First submitted 2010-03-18; First posted 2010-04-02 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Bronchiolitis; Infection; Nitric Oxide
Keywords: RSV Bronchiolitis; Lower Respiratory Viral infection; Exhaled Nitric Oxide
MeSH Terms: conditions — Bronchiolitis; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Exhaled air for Nitric Oxide measurement
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- RSV positive subjects: Subjects admitted to Winthrop University Hospital with lower viral respiratory infection and RSV positive status by DFA and/or Viral culture
- RSV negative subjects: Subjects admitted to Winthrop University Hospital with a lower viral respiratory infection and RSV status negative by DFA and viral culture. these subjects may be positive for other viruses detected by DFA or viral culture (Adenovirus, Influenza A or B, Metapneumovirus or parainfluenza) or not
- Control group: Children in the same age range without respiratory conditions and who are well enough to perform the test from the out patient setting

SUMMARY:
The fraction of exhaled nitric oxide (FeNO) in expired air is a reliable measure of airway inflammation and has been used as a marker in asthma and other respiratory illnesses such as primary ciliary dyskinesia, bronchopulmonary dysplasia (BPD), liver cirrhosis, chronic obstructive pulmonary disease (COPD), cystic fibrosis (CF). Although, some exquisite bench research experiments have demonstrated stimulation of nitric oxide production in respiratory epithelial cells infected with RSV, there is a paucity of clinical data regarding levels of feNO in viral respiratory illness and specifically RSV.

The investigators conducted a pilot study from the fall of 2007 until October of 2009, looking at FeNO levels in RSV infected patients and compared it to non-RSV viral infections. The investigators recruited a total of 28 RSV positive and 1 RSV negative subjects, as well as 4 control subjects. The investigators found FeNO values not statistically significant between the study group (the two-tailed p=0.09, considered not quite significant), but there was a trend of higher FeNO values in the non-RSV group when compared to the RSV group. A larger sample may detect a statistically significance between these 2 groups.

Objectives:

i. To determine if the fraction of exhaled nitric oxide (feNO) is elevated in hospitalized pediatric patients with viral lower respiratory illness when compared with normal subjects without respiratory symptoms.

ii. To determine if there is a difference in feNO level between RSV and non-RSV infection in hospitalized pediatric patients with viral lower respiratory illness.

Method of feNO measurement utilized the offline options for preschool children & infants appropriate for age as described in the 2005 Joint Statement of the American Thoracic Society & the European Respiratory Society when discussing tidal breathing techniques with uncontrolled flow rate.

The investigators plan that our sample sizes for the RSV+ and control groups will be, by design, three times as large as the RSV- group. In order to achieve 80% power, the investigators will then require 45 control and 45 RSV+ patients, and 15 RSV- patients

ELIGIBILITY:
Inclusion Criteria:

* Consecutive children admitted to WUH with a diagnosis of bronchiolitis, viral pneumonia or other significant respiratory viral infection
* The control group will include patient within the same age range as the study group who comes to the pediatric office for a well child visit and has none of the exclusion criteria listed below

Exclusion Criteria:

* Subjects who do not meet the diagnosis for bronchiolitis, viral pneumonia or other significant respiratory viral infection; all patients with underlying diagnosis of asthma/RAD, recurrent wheezing, "recurrent bronchiolitis", allergic rhinitis, atopy, any chronic lung disease, hypertension, heart failure, kidney failure receiving or not dialysis, pulmonary hypertension, primary ciliary dyskinesia, bronchiectasis, alveolitis, lung transplant rejection, pulmonary sarcoidosis, chronic cough (i.e. greater four weeks), systemic sclerosis, hypersensitivity, cystic fibrosis, HIV, sickle cell anemia, cardiac pulmonary bypass, liver cirrhosis, alpha-1 anti-trypsin disease and interstitial lung.

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children admitted to Winthrop University Hospital with lower respiratory tract viral illness, bronchiolitis or pneumonia.
  The control group will include children in the same age range without respiratory conditions and who are well enough to perform the test from the out patient setting
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine if the fraction of exhaled nitric oxide (feNO) is elevated in hospitalized pediatric patients with viral lower respiratory illness when compared with normal subjects without respiratory symptoms | 1 year
To determine if there is a difference in feNO level between RSV and non-RSV infection in hospitalized pediatric patients with viral lower respiratory illness | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Quintos-Alagheband, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Baraldi E, de Jongste JC; European Respiratory Society/American Thoracic Society (ERS/ATS) Task Force. Measurement of exhaled nitric oxide in children, 2001. Eur Respir J. 2002 Jul;20(1):223-37. doi: 10.1183/09031936.02.00293102. PMID 12166573
- [Background] Ricciardolo FL, Sterk PJ, Gaston B, Folkerts G. Nitric oxide in health and disease of the respiratory system. Physiol Rev. 2004 Jul;84(3):731-65. doi: 10.1152/physrev.00034.2003. PMID 15269335
- [Background] Kao YJ, Piedra PA, Larsen GL, Colasurdo GN. Induction and regulation of nitric oxide synthase in airway epithelial cells by respiratory syncytial virus. Am J Respir Crit Care Med. 2001 Feb;163(2):532-9. doi: 10.1164/ajrccm.163.2.9912068. PMID 11179135
- [Background] Beilman G. Exhaled nitric oxide in pathophysiologic states: the substance behind the gas. Chest. 2004 Jan;125(1):11-3. doi: 10.1378/chest.125.1.11. No abstract available. PMID 14718413
- [Background] Baraldi E, Dario C, Ongaro R, Scollo M, Azzolin NM, Panza N, Paganini N, Zacchello F. Exhaled nitric oxide concentrations during treatment of wheezing exacerbation in infants and young children. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1284-8. doi: 10.1164/ajrccm.159.4.9807084. PMID 10194178
- [Background] Gabriele C, Nieuwhof EM, Van Der Wiel EC, Hofhuis W, Moll HA, Merkus PJ, De Jongste JC. Exhaled nitric oxide differentiates airway diseases in the first two years of life. Pediatr Res. 2006 Oct;60(4):461-5. doi: 10.1203/01.pdr.0000238242.39881.64. Epub 2006 Aug 28. PMID 16940253
- [Background] Baraldi E, Ghiro L, Piovan V, Carraro S, Ciabattoni G, Barnes PJ, Montuschi P. Increased exhaled 8-isoprostane in childhood asthma. Chest. 2003 Jul;124(1):25-31. doi: 10.1378/chest.124.1.25. PMID 12853498
- [Background] Jartti T, Makela MJ, Vanto T, Ruuskanen O. The link between bronchiolitis and asthma. Infect Dis Clin North Am. 2005 Sep;19(3):667-89. doi: 10.1016/j.idc.2005.05.010. PMID 16102655
- [Background] Mansbach JM, Camargo CA Jr. Respiratory viruses in bronchiolitis and their link to recurrent wheezing and asthma. Clin Lab Med. 2009 Dec;29(4):741-55. doi: 10.1016/j.cll.2009.07.011. PMID 19892232
- [Background] Sigurs N, Bjarnason R, Sigurbergsson F, Kjellman B. Respiratory syncytial virus bronchiolitis in infancy is an important risk factor for asthma and allergy at age 7. Am J Respir Crit Care Med. 2000 May;161(5):1501-7. doi: 10.1164/ajrccm.161.5.9906076. PMID 10806145
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806